CLINICAL TRIAL: NCT00426244
Title: Osteopathic Manipulative Medicine in Pregnancy: Physiologic and Clinical Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); American Osteopathic Association (Other); American Academy of Osteopathy (Other); Med Ed Foundation of the Am Coll of Osteopathic Obstetricians & Gynecologists (Unknown); Osteopathic Heritage Foundations (Other)
Responsible Party: Principal Investigator, Kendi Hensel, DO, PhD, Associate Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: K23AT003304-01A1 (NIH); 5K23AT003304-05 (NIH)
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Low Back Pain; Pregnancy
Keywords: Osteopathic Manipulative Medicine; Osteopathic Manipulative Treatment; Pregnancy; Physiologic; Gait; Low back pain; Heart rate variability
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Ultrasound (Sham Comparator): In addition to controlling for physician attention during the treatment visit, the SUT used a nonfunctional ultrasound therapy unit that was modified for research purposes to provide both visible and auditory cues that could potentially elicit a placebo response. The physician provided the SUT by placing the applicator head over the subject's clothing and applying sufficient pressure for tactile stimulation of the skin and underlying tissues in the same anatomical distributions as would generally be addressed if the subject were being treated with OMT.
  The subjects assigned to the UOBC only group did not receive any study treatments beyond conventional obstetrical care; however, they were expected to complete data collection forms on the same schedule as all other trial subjects.
  Interventions: Other: Placebo Ultrasound
- Osteopathic Manipulative Treatment (Active Comparator): OMT is a complementary and alternative body-based treatment method in which the patient is evaluated and treated including the musculoskeletal system to improve physiologic functioning and remove impediments to optimal health and functioning.
  Interventions: Other: Osteopathic Manipulative Treatment
- Standard Care (No Intervention): Subject only receives care from her OB provider. Subjects were allowed to receive conventional obstetrical care with the exception of OMT, massage therapy, physical therapy, chiropractic manipulation, or therapeutic ultrasound intended to treat musculoskeletal disorders.

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — OMT is a complementary and alternative body-based treatment method in which the patient is evaluated and treated including the musculoskeletal system to improve physiologic functioning and remove impediments to optimal health and functioning.
  Arms: Osteopathic Manipulative Treatment
Other: Placebo Ultrasound — In addition to controlling for physician attention during the treatment visit, the SUT used a nonfunctional ultrasound therapy unit that was modified for research purposes to provide both visible and auditory cues that could potentially elicit a placebo response. The physician provided the SUT by placing the applicator head over the subject's clothing and applying sufficient pressure for tactile stimulation of the skin and underlying tissues in the same anatomical distributions as would generally be addressed if the subject were being treated with OMT.
  The subjects assigned to the UOBC only group did not receive any study treatments beyond conventional obstetrical care; however, they were expected to complete data collection forms on the same schedule as all other trial subjects.
  Other Names: Sham Ultrasound Therapy
  Arms: Placebo Ultrasound

SUMMARY:
The purpose of this study is to determine to what extent and by what physiological mechanisms Osteopathic Manipulative Medicine (OMM) affects selected conditions related to pregnancy, labor and delivery.

DETAILED DESCRIPTION:
The osteopathic philosophy of health is built on a model in which basic body functions are coordinated and integrated by the musculoskeletal system. Osteopathic medical students are taught to consider these aspects in assessing, diagnosing, and treating the individual patient. As a treatment method that reflects the osteopathic philosophy, osteopathic manipulative medicine (OMM) is a body-based modality in which the patient is evaluated and treated as a whole to improve physiologic functioning and remove impediments to optimal health and functioning.

During pregnancy, a woman's body is challenged by significant and extensive physiological and biomechanical changes. Some physiological changes, such as increased fluid volume and sympathetic tone, may lead to consequences such as edema, preterm labor, and meconium-staining of the amniotic fluid. The biomechanical state of the woman's body is also drastically affected; as the fetus grows and the uterus expands, the center of gravity shifts forward, rotating the pelvis anteriorly and increasing the lordosis of the low back, and may also affect the motion of the hips and legs. These postural changes also have consequences such as low back pain, decreased functional status, and altered gait. Both these physiologic and biomechanical consequences can have a significant long-term impact on the health of the mother and child.

OMM is theorized to facilitate the body's adjustment to the physiological and biomechanical demands of pregnancy and improve the outcomes of pregnancy, labor and delivery. Clinical case studies report reduced back pain, shorter labor, and fewer incidences of peripartum complications in patients who receive prenatal OMM. However, to date we have found no published systematic investigations of the efficacy of OMM in managing the adverse effects that pregnancy has on a woman's musculoskeletal system, nor have we found any published systematic studies to prove the mechanisms of action of OMM in managing pain, edema, or gait in pregnant patients.

Thus, the overall question that guides this proposal is: to what extent and by what physiological mechanisms does Osteopathic Manipulative Medicine (OMM) affect selected conditions related to pregnancy, labor and delivery? Based on the principles and theories of OMM and the limited previous studies, the hypothesis of this study is that OMM improves clinical outcomes including low back pain, functional status, incidence of meconium-stained amniotic fluid, and complications of labor and delivery, and that the physiological changes related to improved autonomic regulation, peripheral hemodynamic regulation, and biomechanical changes related to gait are, in part, responsible for these clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* The woman must have medical clearance from her obstetrician at each study visit
* Must be less than or at 30 weeks gestation at the start of the study

Exclusion Criteria:

* Deemed high risk by the obstetrician (including but not limited to: abruptio placenta, placenta previa, severe pre-eclampsia/eclampsia, vaginal bleeding, gestational diabetes)
* Age 17 years or younger. Females 17 years of age and younger are considered pediatric high risk pregnancies and therefore ineligible for inclusion
* If a patient receives any other manual therapies such as massage, physical therapy, or chiropractic therapy, during the trial, she will be dropped from the study
* Subjects with a history of syncope either before or during this pregnancy will be excluded from participation in the substudy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2006-04; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Low Back Pain and Disability Questionnaire at each visit. | 5 years
Quadruple Visual Analog Scale at each visit. | 5 years
Ware's Short Form-12 (SF-12)at each visit. | 5 years
PHYSIOLOGICAL STUDY -All measures at visit 1 (30 weeks) and visit 4 (36 weeks) | 5 years
Heart rate and blood pressure variability as measured by ECG and power spectral analysis. | 5 years
BIOMECHANICAL STUDY - All measures taken at visit 1 (30 weeks) and visit 4 (36 weeks) | 5 years
Step length as measured by the GAITRite walkway. | 5 years
Foot angle of progression as measured by the GAITRite walkway. | 5 years
Gait Symmetry as measured by the GAITRite walkway. | 5 years

SECONDARY OUTCOMES:
CLINICAL STUDY | 5 years
Subject Confidence in Treatment Assessment at visits 1,7,and 9. | 5 yers
Meconium staining of the amniotic fluid as recorded on the delivery record. | 5 years
Other outcomes of pregnancy, labor and delivery including incidence of high-risk status, incidence of pre-term labor, length of labor, use of forceps or suction device, and pain medication use as recorded in the prenatal and delivery record. | 5 years
PHYSIOLOGICAL STUDY-All measures at visit 1 (30 weeks) and visit 4 (36 weeks) | 5 years
Heart rate as measured by ECG. | 5 years
Arterial pressure as measured by finger photoplethysmographic monitor. | 5 years
Respiration as measured by a strain gauge belt. | 5 years
Saphenous vein diameter and flow as measured by surface ultrasound. | 5 years
Calf muscle EMG as measured by surface electromyographic activity of the gastrocnemius | 5 years
Total leg volume as estimated by strain gauge plethysmography. | 5 years
Tissue water content as measured by surface dielectric probe. | 5 years
Venous flow rate as measured by calf plethysmography. | 5 years
BIOMECHANICAL STUDY -All measures taken at visit 1 (30 weeks) and visit 4 (36 weeks) | 5 years
Gait cadence as measured by the GAITRite walkway. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kendi Hensel, D.O., Ph.D., Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

REFERENCES:
- [Background] Kristiansson P, Svardsudd K, von Schoultz B. Back pain during pregnancy: a prospective study. Spine (Phila Pa 1976). 1996 Mar 15;21(6):702-9. doi: 10.1097/00007632-199603150-00008. PMID 8882692
- [Background] Franklin ME, Conner-Kerr T. An analysis of posture and back pain in the first and third trimesters of pregnancy. J Orthop Sports Phys Ther. 1998 Sep;28(3):133-8. doi: 10.2519/jospt.1998.28.3.133. PMID 9742469
- [Background] Kristiansson P, Svardsudd K, von Schoultz B. Serum relaxin, symphyseal pain, and back pain during pregnancy. Am J Obstet Gynecol. 1996 Nov;175(5):1342-7. doi: 10.1016/s0002-9378(96)70052-2. PMID 8942512
- [Background] Daly JM, Frame PS, Rapoza PA. Sacroiliac subluxation: a common, treatable cause of low-back pain in pregnancy. Fam Pract Res J. 1991 Jun;11(2):149-59. PMID 1829312
- [Background] Lynch FW. The pelvic articulations during pregnancy, labor and the puerperium: An X-ray study. Surgery, Gynecology, and Obstetrics 30: 575-580, 1920.
- [Background] Ostgaard HC, Andersson GB, Schultz AB, Miller JA. Influence of some biomechanical factors on low-back pain in pregnancy. Spine (Phila Pa 1976). 1993 Jan;18(1):61-5. doi: 10.1097/00007632-199301000-00010. PMID 8434326
- [Background] Treadwell RC, Magnus WW. Sacral shear: Review and a new treatment method for obstetricial patients. AAO Journal (Spring): 16-18, 1996.
- [Background] Perkins J, Hammer RL, Loubert PV. Identification and management of pregnancy-related low back pain. J Nurse Midwifery. 1998 Sep-Oct;43(5):331-40. doi: 10.1016/s0091-2182(98)00032-9. PMID 9803711
- [Background] Heckman JD, Sassard R. Musculoskeletal considerations in pregnancy. J Bone Joint Surg Am. 1994 Nov;76(11):1720-30. doi: 10.2106/00004623-199411000-00018. No abstract available. PMID 7962034
- [Background] McIntyre IN, Broadhurst NA. Effective treatment of low back pain in pregnancy. Aust Fam Physician. 1996 Sep;25(9 Suppl 2):S65-7. PMID 8854409
- [Background] Brandy RE, Rottman J, Kappler RE, Veith EK. Forty first Annual AOA Research Conference Abstracts, 1997: Part 1: Osteopathic Manipulation to Treat Musculoskeletal Pain Associated with Pregnancy. JAOA 97(8): 479, 1997.
- [Background] Diakow PR, Gadsby TA, Gadsby JB, Gleddie JG, Leprich DJ, Scales AM. Back pain during pregnancy and labor. J Manipulative Physiol Ther. 1991 Feb;14(2):116-8. PMID 1826921
- [Background] Licciardone JC, Stoll ST, Fulda KG, Russo DP, Siu J, Winn W, Swift J Jr. Osteopathic manipulative treatment for chronic low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1355-62. doi: 10.1097/01.BRS.0000067110.61471.7D. PMID 12838090
- [Background] Andersson GB, Lucente T, Davis AM, Kappler RE, Lipton JA, Leurgans S. A comparison of osteopathic spinal manipulation with standard care for patients with low back pain. N Engl J Med. 1999 Nov 4;341(19):1426-31. doi: 10.1056/NEJM199911043411903. PMID 10547405
- [Background] MacDonald RS, Bell CM. An open controlled assessment of osteopathic manipulation in nonspecific low-back pain. Spine (Phila Pa 1976). 1990 May;15(5):364-70. doi: 10.1097/00007632-199005000-00005. PMID 2141951
- [Background] Koes BW, Assendelft WJ, van der Heijden GJ, Bouter LM. Spinal manipulation for low back pain. An updated systematic review of randomized clinical trials. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2860-71; discussion 2872-3. doi: 10.1097/00007632-199612150-00013. PMID 9112710
- [Background] Cherkin DC, Sherman KJ, Deyo RA, Shekelle PG. A review of the evidence for the effectiveness, safety, and cost of acupuncture, massage therapy, and spinal manipulation for back pain. Ann Intern Med. 2003 Jun 3;138(11):898-906. doi: 10.7326/0003-4819-138-11-200306030-00011. PMID 12779300
- [Background] Wang SM, Dezinno P, Maranets I, Berman MR, Caldwell-Andrews AA, Kain ZN. Low back pain during pregnancy: prevalence, risk factors, and outcomes. Obstet Gynecol. 2004 Jul;104(1):65-70. doi: 10.1097/01.AOG.0000129403.54061.0e. PMID 15229002
- [Background] Cleary GM, Wiswell TE. Meconium-stained amniotic fluid and the meconium aspiration syndrome. An update. Pediatr Clin North Am. 1998 Jun;45(3):511-29. doi: 10.1016/s0031-3955(05)70025-0. PMID 9653434
- [Background] March of Dimes. Prenatal Overview: PeriStats (2005). Retrieved January 21, 2005, from www.marchofdimes.com/peristats.
- [Background] Klingner MC, Kruse J. Meconium aspiration syndrome: pathophysiology and prevention. J Am Board Fam Pract. 1999 Nov-Dec;12(6):450-66. doi: 10.3122/jabfm.12.6.450. PMID 10612363
- [Background] King HH, Tettambel MA, Lockwood MD, Johnson KH, Arsenault DA, Quist R. Osteopathic manipulative treatment in prenatal care: a retrospective case control design study. J Am Osteopath Assoc. 2003 Dec;103(12):577-82. PMID 14740980
- [Background] Whiting LM. Can the Length of Labor be Shortened by Osteopathic Treatment. Journal of the American Osteopathic Association (11): 917-921, 1911.
- [Background] Whiting LM. The osteopathic management of pregnancy and the reduction of obstetrical mortality. Journal of the American Osteopathic Association 33(8): 531-533, 1934.
- [Background] Still, EM. Osteopathic Obstetrics. Journal of Osteopathy 4(4): 203-204, 1897.
- [Background] Dooley W. Osteopathy's Contribution to Prenatal Care. Journal of the American Osteopathic Association 46(1): 6-7, 1946.
- [Background] Guthrie RA, Martin RH. Effect of pressure applied to the upper thoracic (placebo) versus lumbar areas (osteopathic manipulative treatment) for inhibition of lumbar myalgia during labor. J Am Osteopath Assoc. 1982 Dec;82(4):247-51. No abstract available. PMID 6218150
- [Background] Guthrie RA. Lumbar inhibitory pressure for lumbar myalgia during contractions of the gravid uterus at term. J Am Osteopath Assoc. 1980 Dec;80(4):264-6. No abstract available. PMID 6453858
- [Background] Hart LM. Obstetrical practice. Journal of American Osteopathic Association (July): 609-614, 1918.
- [Background] King HH, Osteopathic manipulative treatment in prenatal care: Evidence supporting improved outcomes and health policy implications. The American Academy of Osteopathy Journal (Summer): 25-33, 2000.
- [Background] TAYLOR GW. The osteopathic management of nausea and vomiting of pregnancy. J Am Osteopath Assoc. 1949 Jul;48(11):581. No abstract available. PMID 18152732
- [Background] Troyanovich S. Pregnancy and the Chiropractic Advantage. Today's Chiropractic, 21(6): 46-48, 1992.
- [Background] Laman J, King M. Promoting healthy babies. NCSL Legisbrief National Conference of State Legislatures. February 1994.
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Greenwood JP, Stoker JB, Walker JJ, Mary DA. Sympathetic nerve discharge in normal pregnancy and pregnancy-induced hypertension. J Hypertens. 1998 May;16(5):617-24. doi: 10.1097/00004872-199816050-00009. PMID 9797173
- [Background] McLean M, Smith R. Corticotrophin-releasing hormone and human parturition. Reproduction. 2001 Apr;121(4):493-501. doi: 10.1530/rep.0.1210493. PMID 11277868
- [Background] Hobel C, Culhane J. Role of psychosocial and nutritional stress on poor pregnancy outcome. J Nutr. 2003 May;133(5 Suppl 2):1709S-1717S. doi: 10.1093/jn/133.5.1709S. PMID 12730488
- [Background] Current Obstetric & Gynecologic Diagnosis & Treatment, 8th Edition. Cardiovasvular System. Chapter 7, 150-154.
- [Background] Kuchera ML, Kuchera WA. (1994).Osteopathic Considerations in Systemic Dysfunction, revised 2nd Ed. Greyden Press; Columbus, OH; pp 55, 85, 187, 193.
- [Background] Smutny CJ, Wells WR, Bosak A. Osteopathic Considerations in Parkinson's Disease. Journal of the American Osteopathic Association 98 (7): 389, 1998.
- [Background] Wells MR, Giantinoto S, D'Agate D, Areman RD, Fazzini EA, Dowling D, Bosak A. Standard osteopathic manipulative treatment acutely improves gait performance in patients with Parkinson's disease. J Am Osteopath Assoc. 1999 Feb;99(2):92-8. doi: 10.7556/jaoa.1999.99.2.92. PMID 10079641
- [Background] Wells MR, McCarty CL, Smutny CJ, Scandalis TA, Dittrich F, Fazzini EA Osteopathic Manipulation in the Management of Parkinson's Disease: Preliminary Findings. The Journal of the American Osteopathic Association 100(8): 522, 2000.
- [Background] Guadagnino MR. Spinal manipulative therapy for 12 pregnant patients suffering from low back pain. Journal of Chiropractic Technique 11(3): 108-112, 1999.
- [Background] Smith ML, Raven PB. Cardiovascular responses to lower body negative pressure in endurance and static exercise-trained men. Med Sci Sports Exerc. 1986 Oct;18(5):545-50. PMID 3773671
- [Background] Carter R 3rd, Watenpaugh DE, Wasmund WL, Wasmund SL, Smith ML. Muscle pump and central command during recovery from exercise in humans. J Appl Physiol (1985). 1999 Oct;87(4):1463-9. doi: 10.1152/jappl.1999.87.4.1463. PMID 10517779
- [Background] Ogoh S, Volianitis S, Nissen P, Wray DW, Secher NH, Raven PB. Carotid baroreflex responsiveness to head-up tilt-induced central hypovolaemia: effect of aerobic fitness. J Physiol. 2003 Sep 1;551(Pt 2):601-8. doi: 10.1113/jphysiol.2003.046029. Epub 2003 Jun 17. PMID 12813144
- [Background] Yoshiuchi K, Quigley KS, Ohashi K, Yamamoto Y, Natelson BH. Use of time-frequency analysis to investigate temporal patterns of cardiac autonomic response during head-up tilt in chronic fatigue syndrome. Auton Neurosci. 2004 Jun 30;113(1-2):55-62. doi: 10.1016/j.autneu.2004.05.001. PMID 15296795
- [Background] Butler GC, Yamamoto Y, Xing HC, Northey DR, Hughson RL. Probing heart rate and blood pressure control mechanisms during graded levels of lower body negative pressure (LBNP). Microgravity Q. 1992 Apr;2(2):133-40. PMID 11541049
- [Background] Webster KE, Wittwer JE, Feller JA. Validity of the GAITRite walkway system for the measurement of averaged and individual step parameters of gait. Gait Posture. 2005 Dec;22(4):317-21. doi: 10.1016/j.gaitpost.2004.10.005. Epub 2004 Dec 10. PMID 16274913
- [Background] Hitchcock ME. Osteopathic Care in Pregnancy. Osteopathic Annals (December): 19-30, 1976.
- [Background] Graham KE, Shaw HH, Mills M, Cotton L. Pregnancy, 3rd Trimester and Pre-Delivery: Goals of OMM in Pregnant Patient during Third Trimester and Pre-Delivery. Anatomic and Physiologic Basis of Osteopathic Manipulative Medicine in Visceral Disease. 1st Edition, 74-75, 2001.
- [Background] Stiles EG. Osteopathic manipulation in a hospital environment. J Am Osteopath Assoc. 1976 Dec;76(4):243-58. No abstract available. PMID 1049598
- [Background] Berg G, Hammar M, Moller-Nielsen J, Linden U, Thorblad J. Low back pain during pregnancy. Obstet Gynecol. 1988 Jan;71(1):71-5. PMID 2962023
- [Background] Price DD, Harkins SW. Psychophysical Approaches to Pain Measurement and Assessment. In Turk DC, Melzack R, Editors: Handbook of Pain Assessment, New York: Guliford Press, 1992: 11-132.
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Stratford PW, Binkley J, Solomon P, Gill C, Finch E. Assessing change over time in patients with low back pain. Phys Ther. 1994 Jun;74(6):528-33. doi: 10.1093/ptj/74.6.528. PMID 8197239
- [Background] Beurskens AJHM, de Vet HCW, Koke AJA. Responsiveness of functional status in low back pain: a comparison of different instruments. Pain. 1996 Apr;65(1):71-76. doi: 10.1016/0304-3959(95)00149-2. PMID 8826492
- [Background] Parati G, Saul JP, Di Rienzo M, Mancia G. Spectral analysis of blood pressure and heart rate variability in evaluating cardiovascular regulation. A critical appraisal. Hypertension. 1995 Jun;25(6):1276-86. doi: 10.1161/01.hyp.25.6.1276. PMID 7768574
- [Background] Pagani M, Lombardi F, Guzzetti S, Rimoldi O, Furlan R, Pizzinelli P, Sandrone G, Malfatto G, Dell'Orto S, Piccaluga E, et al. Power spectral analysis of heart rate and arterial pressure variabilities as a marker of sympatho-vagal interaction in man and conscious dog. Circ Res. 1986 Aug;59(2):178-93. doi: 10.1161/01.res.59.2.178. PMID 2874900
- [Background] Malliani A, Lombardi F, Pagani M. Power spectrum analysis of heart rate variability: a tool to explore neural regulatory mechanisms. Br Heart J. 1994 Jan;71(1):1-2. doi: 10.1136/hrt.71.1.1. No abstract available. PMID 8297682
- [Background] Gotshall RW, Davrath LR. Bioelectric impedance as an index of thoracic fluid. Aviat Space Environ Med. 1999 Jan;70(1):58-61. PMID 9895022
- [Background] Johnson JM. Exercise and the cutaneous circulation. Exerc Sport Sci Rev. 1992;20:59-97. PMID 1623893
- [Background] Nuutinen J, Lahtinen T, Turunen M, Alanen E, Tenhunen M, Usenius T, Kolle R. A dielectric method for measuring early and late reactions in irradiated human skin. Radiother Oncol. 1998 Jun;47(3):249-54. doi: 10.1016/s0167-8140(97)00234-x. PMID 9681887
- [Background] Nuutinen J, Ikaheimo R, Lahtinen T. Validation of a new dielectric device to assess changes of tissue water in skin and subcutaneous fat. Physiol Meas. 2004 Apr;25(2):447-54. doi: 10.1088/0967-3334/25/2/004. PMID 15132310
- [Background] Gamble J, Joyner MJ, Dietz NM, Shepherd JT. A restrospective perspective. J Appl Physiol (1985). 2005 Feb;98(2):762; author reply 762-3. doi: 10.1152/japplphysiol.00773.2004. PMID 15649884
- [Background] Welsch MA, Alomari M, Parish TR, Wood RH, Kalb D. Influence of venous function on exercise tolerance in chronic heart failure. J Cardiopulm Rehabil. 2002 Sep-Oct;22(5):321-6. doi: 10.1097/00008483-200209000-00002. PMID 12370591
- [Background] Johnson K. An Integrated Approach for Treating the OB Patient: Treating the Five Diaphrams of the Body, Part I. American Academy of Osteopathy Journal (Winter): 6-9, 1991.
- [Background] Schobel HP, Fischer T, Heuszer K, Geiger H, Schmieder RE. Preeclampsia -- a state of sympathetic overactivity. N Engl J Med. 1996 Nov 14;335(20):1480-5. doi: 10.1056/NEJM199611143352002. PMID 8890098
- [Background] Ware JE, Kosinski M, Dewey JE. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: QualityMetric Incorporated, 2000.
- [Derived] Hensel KL, Roane BM, Chaphekar AV, Smith-Barbaro P. PROMOTE Study: Safety of Osteopathic Manipulative Treatment During the Third Trimester by Labor and Delivery Outcomes. J Am Osteopath Assoc. 2016 Nov 1;116(11):698-703. doi: 10.7556/jaoa.2016.140. PMID 27802555